CLINICAL TRIAL: NCT03060408
Title: Comparison of Intraoperative Basal Fluid Requirements in Distal Pancreatectomy - Laparotomy vs. Laparoscopy: A Retrospective Cohort Study
Brief Title: Comparison of Fluid Requirements in Pancreatectomy: Laparotomy vs. Laparoscopy
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, Principal Investigator, Resident of Anesthesiology and Pain medicine, Seoul National University Bundang Hospital
Other Study IDs: B-1508-312-102
Record Dates: First submitted 2017-01-31; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pancreatectomy; Fluid Therapy; Laparoscopy
Keywords: Fluid Therapy; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Open: Patients underwent open distal pancreatectomy
- Laparoscopic: Patients underwent laparoscopic distal pancreatectomy

SUMMARY:
In this retrospective cohort study, the investigators reviewed and analyzed the electronic medical records of consecutive patients who underwent distal pancreatectomy either via laparotomy or laparoscopy. Intraoperative fluid administration amount, postoperative complications, length of hospital stay, and readmission rate were evaluated. The total fluid amounts were calculated using the sum of colloids multiplied by 1.5 or 2.0 and crystalloids.

DETAILED DESCRIPTION:
There has been recent progress in intraoperative fluid therapy. However, little is known about intraoperative fluid therapy in laparoscopic surgery. The purpose of this study is to determine whether there are differences in the basal fluid requirements during surgery between laparotomy and laparoscopic distal pancreatectomy. This study analyzed the records between June 2006 and March 2016. And 253 patients who underwent distal pancreatectomy via either laparotomy (73 patients) or laparoscopy (180 patients). This study was based on a retrospective review and analysis of the electronic medical records. The volume of intraoperative fluid administered, postoperative complications, length of hospital stay, and readmission rate were evaluated. The total volume of fluids was calculated as the sum of the volume of crystalloid plus the volume of colloid multiplied by 1.5 or 2.0.

ELIGIBILITY:
Inclusion Criteria:

* indication of distal pancreatectomy

Exclusion Criteria:

* transfusion
* ASA physical status over 4
* co-operate other surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: indication of distal pancreatectomy
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
intraoperatively administered fluid amounts | one year